CLINICAL TRIAL: NCT03021694
Title: Testing of Micellar Casein, Blended Micellar Casein and Native Whey, Versus Native Whey to Determine Post-ingestion Aminoacidemia, Glycemia, and Insulinemia in Young Adult Men
Brief Title: Testing of Micellar Casein, Blended Micellar Casein and Native Whey
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Stuart Phillips, Professor, McMaster University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Aminoacidemia_Whey/Casein
Record Dates: First submitted 2017-01-11; First posted 2017-01-16 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Dietary Modification
MeSH Terms: interventions — Blood Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Young Males Week 1 (Experimental): Six separate 3 x 14 [condition (micellar casein, micellar casein and native whey blend, and native whey) x time (-15min, 0 min, 15min, 30min, 45min, 60min, 90min, 150min, 180min, 210min, 240min, 270min, 300min, and 360min)] repeated measures ANOVAs will be used to analyze blood concentrations of leucine, ∑branched chain amino acids, ∑essential amino acids, ∑amino acids, glucose, and insulin.
  Interventions: Dietary Supplement: Testing of micellar casein, blended micellar casein and native whey, versus native whey to determine post-ingestion aminoacidemia, glycemia, and insulinemia in young adult men
- Young Males Week 3 (Experimental): Six separate 3 x 14 [condition (micellar casein, micellar casein and native whey blend, and native whey) x time (-15min, 0 min, 15min, 30min, 45min, 60min, 90min, 150min, 180min, 210min, 240min, 270min, 300min, and 360min)] repeated measures ANOVAs will be used to analyze blood concentrations of leucine, ∑branched chain amino acids, ∑essential amino acids, ∑amino acids, glucose, and insulin.
  Interventions: Dietary Supplement: Testing of micellar casein, blended micellar casein and native whey, versus native whey to determine post-ingestion aminoacidemia, glycemia, and insulinemia in young adult men
- Young Males Week 5 (Experimental): Six separate 3 x 14 [condition (micellar casein, micellar casein and native whey blend, and native whey) x time (-15min, 0 min, 15min, 30min, 45min, 60min, 90min, 150min, 180min, 210min, 240min, 270min, 300min, and 360min)] repeated measures ANOVAs will be used to analyze blood concentrations of leucine, ∑branched chain amino acids, ∑essential amino acids, ∑amino acids, glucose, and insulin.
  Interventions: Dietary Supplement: Testing of micellar casein, blended micellar casein and native whey, versus native whey to determine post-ingestion aminoacidemia, glycemia, and insulinemia in young adult men

INTERVENTIONS:
Dietary Supplement: Testing of micellar casein, blended micellar casein and native whey, versus native whey to determine post-ingestion aminoacidemia, glycemia, and insulinemia in young adult men

SUMMARY:
The importance of protein in nutrition is momentous to ones health. Dietary proteins are essentially nutritional because they contain amino acids, which the body uses to build its own proteins, as well as other molecules that are essential for life. Protein when consumed, travels through your digestive system and is absorbed. They then enter the blood for transport to bodily tissues, and therefore, can be detected by blood sampling. There are differing amounts of each amino acid found in different types of protein supplements. Certain amino acids (the essential amino acids) are helping in stimulating muscle growth and helping to maintain muscle mass and function. It is important to understand how quickly these amino acids can be detected in your blood as well as how they affect blood glucose (blood sugar) and insulin activity. Understanding the effects of protein type on changes in levels of blood amino acids, glucose and insulin will provide helpful insight for the suggestion of supplement use.

DETAILED DESCRIPTION:
The importance of protein in nutrition is momentous to ones health. Dietary proteins are essentially nutritional because of their constituent amino acids, which the body uses to synthesize its own proteins, as well as nitrogen-containing molecules that are essential for life. The Recommended Dietary Allowance (RDA) for daily protein intake in healthy adults is 0.8 g/kgBW/day. Younger individuals who participate in recreational or competitive activities, however, often attempt to go beyond the RDA by using protein supplements to help increase performance. For example, it was demonstrated that protein supplementation in conjunction with an eight-week resistance-training program elicited greater improvements in muscle hypertrophy and strength when compared to carbohydrate supplementation in untrained men. There were 3.2 to 17.5% increases in muscle cross-sectional area of the quadriceps femoris musculature and 14.5 to 30.3% strength gains in the leg extensors. Furthermore, several expert groups have recently advocated that certain individuals, such as older persons, should increase their daily intake to 1.0 to 1.5 g/kgBW/day to support the preservation of muscle and function. Other conditions also place greater than normal demands on amino acids, such as hypercatabolic stressed states, like that experienced by burn patients who's muscle protein breakdown rate increases by impairment to inward transmembrane transport of circulating blood amino acids. It was also found that an experimental enriched protein "medical food" comprised of 27% of calories as total protein resulted in postprandial increases in MPS rates for 5 hours by ∼33% (0.073 ± 0.023%∙h-1 to 0.097 ± 0.033%∙h-1) in advanced cancer patients. Thus, continually reassessing new and innovative nutrient therapies is necessary for extending the findings of existing studies after technological advances, and for providing nutritional support-to-support health.

It is well known that dietary protein is a powerful transient stimulator of the muscle protein synthetic rate (MPS) whereby changes in MPS in response to feeding may be regulated by specific downstream target proteins of mammalian target of rapamycin signaling, such as S6K1, rpS6, and eIF2B. A meal deficient in protein, however, does not increase the rate of MPS because a rise in the bioavailability of amino acids does not occur. In addition, the source of dietary proteins has been shown to impact postprandial blood levels of amino acids. The concept that certain types of proteins are "fast acting" or "slow acting" has been shown to affect the postprandial profile of amino acids appearing in the systemic circulation. Native whey and micellar casein are both dairy proteins that contain a similar amount of essential (EAA), but blood EAA levels increase faster and to a higher level after the consumption of whey protein. Differences in gastric emptying, digestion and absorption kinetics between micellar casein and native whey are suggested to be the underlying factors. Nonetheless, micellar casein protein has been shown to protract MPS in humans. Despite the significant amount of information gained with respect to both of these protein sources, the effects of combinatorial formulations on the postprandial profile of amino acids appearing in the blood is less well known. The purpose of the present study is to test a novel blend of micellar casein combined with native whey to determine post-ingestion aminoacidemia, glycemia, and insulinemia in young adult men.

ELIGIBILITY:
Inclusion Criteria:

* 10 participants will be included in this study.
* Each participant will consume only one of the supplements in a double-blinded fashion during three separate visits and there will be approximately 1 week between each visit.
* In order to participate in this study, each participant must be male, between the ages of 18 and 30 years (inclusive) and cannot be a smoker or user of tobacco products.

Exclusion Criteria:

* The exclusion requirements for this study include the following conditions:

  * Take any analgesic or anti-inflammatory drugs(s), prescription or non-prescription, chronically will be excluded. However, a washout period of 4 weeks will be suitable for participation.
  * A history of neuromuscular problems or muscle and/or bone wasting diseases
  * Any acute or chronic illness, cardiac, pulmonary, liver, or kidney abnormalities, uncontrolled hypertension, insulin- or non-insulin dependent diabetes or other metabolic disorders-all ascertained through medical history screening questionnaires
  * Use medications known to affect protein metabolism (i.e. corticosteroids, non-steroidal anti-inflammatories, or prescription strength acne medications)

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2017-09-10 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Postprandial blood amino acid concentrations | 360 minutes
  repeated blood draws
Postprandial blood insulin concentrations | 360 minutes
  repeated blood draws
Postprandial blood glucose concentrations | 360 minutes
  repeated blood draws

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise Metabolism Research Laboratory, McMaster Univeristy, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rand WM, Pellett PL, Young VR. Meta-analysis of nitrogen balance studies for estimating protein requirements in healthy adults. Am J Clin Nutr. 2003 Jan;77(1):109-27. doi: 10.1093/ajcn/77.1.109. PMID 12499330
- [Background] Coburn JW, Housh DJ, Housh TJ, Malek MH, Beck TW, Cramer JT, Johnson GO, Donlin PE. Effects of leucine and whey protein supplementation during eight weeks of unilateral resistance training. J Strength Cond Res. 2006 May;20(2):284-91. doi: 10.1519/R-17925.1. PMID 16686554
- [Background] Bauer JM, Verlaan S, Bautmans I, Brandt K, Donini LM, Maggio M, McMurdo ME, Mets T, Seal C, Wijers SL, Ceda GP, De Vito G, Donders G, Drey M, Greig C, Holmback U, Narici M, McPhee J, Poggiogalle E, Power D, Scafoglieri A, Schultz R, Sieber CC, Cederholm T. Effects of a vitamin D and leucine-enriched whey protein nutritional supplement on measures of sarcopenia in older adults, the PROVIDE study: a randomized, double-blind, placebo-controlled trial. J Am Med Dir Assoc. 2015 Sep 1;16(9):740-7. doi: 10.1016/j.jamda.2015.05.021. Epub 2015 Jul 10. PMID 26170041
- [Background] Deutz NE, Bauer JM, Barazzoni R, Biolo G, Boirie Y, Bosy-Westphal A, Cederholm T, Cruz-Jentoft A, Krznaric Z, Nair KS, Singer P, Teta D, Tipton K, Calder PC. Protein intake and exercise for optimal muscle function with aging: recommendations from the ESPEN Expert Group. Clin Nutr. 2014 Dec;33(6):929-36. doi: 10.1016/j.clnu.2014.04.007. Epub 2014 Apr 24. PMID 24814383
- [Background] Murphy CH, Oikawa SY, Phillips SM. Dietary Protein to Maintain Muscle Mass in Aging: A Case for Per-meal Protein Recommendations. J Frailty Aging. 2016;5(1):49-58. doi: 10.14283/jfa.2016.80. PMID 26980369
- [Background] Biolo G, Fleming RY, Maggi SP, Nguyen TT, Herndon DN, Wolfe RR. Inverse regulation of protein turnover and amino acid transport in skeletal muscle of hypercatabolic patients. J Clin Endocrinol Metab. 2002 Jul;87(7):3378-84. doi: 10.1210/jcem.87.7.8699. PMID 12107253
- [Background] Tisdale MJ. Mechanisms of cancer cachexia. Physiol Rev. 2009 Apr;89(2):381-410. doi: 10.1152/physrev.00016.2008. PMID 19342610
- [Background] Koopman R, Crombach N, Gijsen AP, Walrand S, Fauquant J, Kies AK, Lemosquet S, Saris WH, Boirie Y, van Loon LJ. Ingestion of a protein hydrolysate is accompanied by an accelerated in vivo digestion and absorption rate when compared with its intact protein. Am J Clin Nutr. 2009 Jul;90(1):106-15. doi: 10.3945/ajcn.2009.27474. Epub 2009 May 27. PMID 19474134
- [Background] Moore DR, Robinson MJ, Fry JL, Tang JE, Glover EI, Wilkinson SB, Prior T, Tarnopolsky MA, Phillips SM. Ingested protein dose response of muscle and albumin protein synthesis after resistance exercise in young men. Am J Clin Nutr. 2009 Jan;89(1):161-8. doi: 10.3945/ajcn.2008.26401. Epub 2008 Dec 3. PMID 19056590
- [Background] Katsanos CS, Kobayashi H, Sheffield-Moore M, Aarsland A, Wolfe RR. A high proportion of leucine is required for optimal stimulation of the rate of muscle protein synthesis by essential amino acids in the elderly. Am J Physiol Endocrinol Metab. 2006 Aug;291(2):E381-7. doi: 10.1152/ajpendo.00488.2005. Epub 2006 Feb 28. PMID 16507602
- [Background] Luiking YC, Abrahamse E, Ludwig T, Boirie Y, Verlaan S. Protein type and caloric density of protein supplements modulate postprandial amino acid profile through changes in gastrointestinal behaviour: A randomized trial. Clin Nutr. 2016 Feb;35(1):48-58. doi: 10.1016/j.clnu.2015.02.013. Epub 2015 Mar 5. PMID 25790724
- [Background] Tipton KD, Elliott TA, Cree MG, Wolf SE, Sanford AP, Wolfe RR. Ingestion of casein and whey proteins result in muscle anabolism after resistance exercise. Med Sci Sports Exerc. 2004 Dec;36(12):2073-81. doi: 10.1249/01.mss.0000147582.99810.c5. PMID 15570142
- [Background] Boirie Y, Dangin M, Gachon P, Vasson MP, Maubois JL, Beaufrere B. Slow and fast dietary proteins differently modulate postprandial protein accretion. Proc Natl Acad Sci U S A. 1997 Dec 23;94(26):14930-5. doi: 10.1073/pnas.94.26.14930. PMID 9405716